CLINICAL TRIAL: NCT07163481
Title: A Phase Ib, Open-label, Modular Trial to Evaluate Sacituzumab Govitecan in Combination With Endocrine Therapy in Patients With HR-positive, HER2-negative Metastatic Breast Cancer Progressed on CDK4/6 Inhibitors
Brief Title: A Trial to Evaluate Sacituzumab Govitecan in Combination With Endocrine Therapy in Patients With HR-positive, HER2-negative Metastatic Breast Cancer Progressed on CDK4/6 Inhibitors
Acronym: SoGreat
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-CN-979-6924
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stage IV (Metastatic) Breast Cancer
Keywords: Sacituzumab Govitecan; Breast Neoplasms
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — sacituzumab govitecan; Fulvestrant; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Module 1: Progressed on Aromatase Inhibitors Combined with CDK4/6 Inhibitors (Experimental): Patients Progressed on Aromatase Inhibitors Combined with CDK4/6 Inhibitors
  Intervention:
  Sacituzumab Govitecan 10 mg/kg intravenously on Days 1 and 8 of 21-day cycles Combined with Fulvestrant 500 mg intramuscularly into the buttock on Day 1 of 28-day cycles and Cycle 1 Day 15
  Interventions: Drug: Sacituzumab Govitecan + Fulvestrant
- Module 2: Progressed on Selective Estrogen Receptor Degrader Combined with CDK4/6 Inhibitors (Experimental): Patients Progressed on Selective Estrogen Receptor Degrader Combined with CDK4/6 Inhibitors
  Intervention:
  Sacituzumab Govitecan 10 mg/kg intravenously on Days 1 and 8 of 21-day cycles Combined with one of the two
  Investigator's choice of aromatase inhibitors (ICAI), orally, once daily:
  * Anastrozole 1 mg, or
  * Exemestane 25 mg
  Interventions: Drug: Sacituzumab Govitecan + Anastrozole / Exemestane

INTERVENTIONS:
Drug: Sacituzumab Govitecan + Fulvestrant — Sacituzumab Govitecan 10 mg/kg intravenously on Days 1 and 8 of 21-day cycles Combined with Fulvestrant 500 mg intramuscularly into the buttock on Day 1 of 28-day cycles and Cycle 1 Day 15
  Arms: Module 1: Progressed on Aromatase Inhibitors Combined with CDK4/6 Inhibitors
Drug: Sacituzumab Govitecan + Anastrozole / Exemestane — Sacituzumab Govitecan 10 mg/kg intravenously on Days 1 and 8 of 21-day cycles Combined with One of the Two Investigator's choice of aromatase inhibitors (ICAI), orally, once daily: Anastrozole 1 mg Exemestane 25 mg
  Arms: Module 2: Progressed on Selective Estrogen Receptor Degrader Combined with CDK4/6 Inhibitors

SUMMARY:
SoGreat is an open-label, single-arm, modular, two-stage, Phase Ib/II study. SoGreat (Part 1) is an open-label, modular, Phase Ib study.

DETAILED DESCRIPTION:
SoGreat is an open-label, single-arm, modular, two-stage, Phase Ib/II study. SoGreat (Part 1) is an open-label, modular, Phase Ib study.

The study consisted of an up to 28-day Screening period, followed by the Treatment Phase and Follow-up.

Screen Period:

It is to determine baseline disease characteristics and to confirm patient eligibility prior to randomization and treatment.

If tumor evaluation performed as part of routine clinical practice provides valid results within the permitted time frame (within 28 days prior to C1D1), there is no need to repeat tumor imaging at the screening visit. Bone scan (99m technetium polyphosphate scintigraphy, whole body bone MRI, or 18F-NaF/FDG PET) is required to assess bone metastasis within 6 weeks prior to C1D1 (historical scans are acceptable);

Eligible patients will be assigned to one of the following 2 treatment modules based on different endocrine agents previously combined with CDK4/6 inhibitors in the advanced first-line setting:

Module 1: Fulvestrant 500 mg IM, Days 1 & 15 of cycle 1 and Day 1 for all other cycles thereafter IF patients progressed on the first-line treatment of CDK4/6i combined with aromatase inhibitors.

Module 2: one of the two investigators' choices of aromatase inhibitors (ICAI) oral QD IF patients progressed on the first-line treatment of CDK4/6i combined with Fulvestrant. Mutual substitution is not allowed during the study.

Treatment Phase:

Sacituzumab Govitecan will be administered in 21-day cycles on Days 1 and 8; the next cycle should start 14 days after the Day 8 dose (i.e., the Day 8 infusion will be counted as the first day of that 14-day period). However, visit windows of 1 day prior to and 2 days after the scheduled infusion are permitted. The scheduled Day 1 and Day 8 infusions may be delayed for up to 3 weeks for treatment-related toxicities.

Dose modifications are permitted for sacituzumab govitecan per product inserts (NMPA v2023/03/01).

Dose modifications are NOT permitted for endocrine therapy. Treatment was continued until disease progression, unacceptable toxicity, or patient or physician decision. Patients who have experienced a complete response (CR) were to be treated for a minimum of 12 months and/or until disease progression or unacceptable toxicity, after confirmation of response. Tumor measurements by computed tomography (CT) scan or magnetic resonance imaging (MRI; chest, abdomen, pelvis, other areas of known/suspected involvement, with contrast as appropriate) were to be performed every 6 weeks to determine response to treatment, after Week 12, assessments were to be performed every 12 weeks. The response was evaluated using the RECIST v 1.1. Disease progression per RECIST v 1.1 leading to treatment withdrawal was assessed by the Investigator. Clinical progression leading to patient discontinuation was to be documented also by CT/MRI scan, if possible.

NCI-CTCAE v 5.0 toxicity grades were used to classify safety evaluations and adverse events, including serious adverse events (SAEs). Adverse event reporting was started after written informed consent was obtained from the patient and continued for 30 days after the last administration of the IP.

End of Treatment visit was to be planned within 7 days from the decision to discontinue the investigational product (IP), or before the start of any other antitumor therapy. If the patient discontinues study treatment prematurely without objective progression and initiating any other antitumor therapy, then tumor assessment was to be continued in follow-up visits until progression or death.

Follow-Up:

A safety Follow-up visit was to be performed 30 days (+/- 3 days) after the last administration of IP. Survival follow-up was to be performed every 12 weeks (+/- 1 week) after the Safety Follow-up visit, might be by telephone, and included the documentation of any further active therapy administrated for their breast cancer.

Periodic evaluations of the study data were conducted by a Safety Monitoring Committee (SMC) to ensure patient safety and the validity and scientific merit of the study.

ELIGIBILITY:
Inclusion Criteria:Patients must meet the following criteria at screening:

1. Female or male patients, 18 years of age or older, able to understand and give written informed consent.
2. ECOG performance status of 0 or 1.
3. Men, pre-menopausal or perimenopausal women must use gonadotropin-releasing hormone agonists (such as goserelin) in a standardized manner.
4. Postmenopausal women must meet one of the following criteria:

   1. bilateral oophorectomy.
   2. age 60 years or older.
   3. age <60 years and natural menopause (not induced by medication) for more than 12 months with follicle-stimulating hormone (FSH) and estradiol levels in the postmenopausal range.
5. Histologically documented breast cancer that:

   1. Is locally advanced inoperable or metastatic recurrence.
   2. Is documented as HR-positive, HER2-negative (either ER and/or PgR positive [ER or PgR 1%]; HER2 negative [IHC 2+/ISH-; IHC1+/ISH- or untested; IHC 0/ISH- or untested]) per ASCO/CAP guidelines in the metastatic setting. If a patient has had multiple ER/PgR/HER2 results after metastatic disease, the most recent test result will be used to confirm eligibility.
6. Radiologic or objective evidence of disease progression on or after the last systemic therapy prior to starting study treatment.
7. Must have had disease progression on CDK4/6i combined with endocrine therapy administrated as the first line and the only therapy for metastatic disease. The time till progression (TTP) for the first line CDK4/6 must be no less than 6 months.
8. Patients who received adjuvant endocrine therapy with or without CDK4/6i with curative intent for early breast cancer are eligible, as long as they relapse after the first 24 months of adjuvant endocrine therapy.
9. No prior chemotherapy for advanced or metastatic breast cancer. Patients who have received chemotherapy in the neo-adjuvant or adjuvant setting are eligible, as long as they have had a disease-free interval (defined as completion of systemic chemotherapy to the diagnosis of advanced or metastatic disease) of >12 months.
10. Measurable disease by CT or MRI in accordance with RECIST v 1.1, the bone-only disease was not measurable and was not permitted.
11. Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (hemoglobin ≥ 9 g/dL, ANC ≥ 1500/mm 3 , and platelets ≥ 100,000/µL).
12. Adequate hepatic function (bilirubin ≤ 1.5 × ULN, AST and ALT ≤ 2.5 × ULN or ≤ 5 × ULN if known liver metastases, and serum albumin > 3 g/dL).
13. Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation
14. Recovered from all prior treatment-related toxicities to Grade 1 or less by NCI-CTCAE v 5.0 (except alopecia or peripheral neuropathy, which should be Grade 2 or less).
15. Willing and able to comply with the requirements and restrictions in this protocol.

    -

Exclusion Criteria: Patients must NOT meet the following criteria at screening:

1. Positive serum pregnancy test or women who are breastfeeding.
2. Women of childbearing potential or fertile men unwilling to use highly effective contraception during the study and up to 6 months after treatment discontinuation in women of childbearing potential and 3 months in males post last IP administration.
3. Known hypersensitivity to the study drug, its metabolites, or formulation excipient.
4. Requirement for ongoing therapy with or prior use of any prohibited medications listed in Section 4.2.6.
5. Have had a prior anticancer biologic agent within 4 weeks prior to enrollment or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to enrollment and have not recovered (i.e., ≥ Grade 2 is considered not recovered) from AEs at the time of study entry.
6. Have not recovered (i.e., ≥ Grade 2 is considered not recovered) from AEs due to a previously administered agent.

   * Note: patients with any grade neuropathy or alopecia are an exception to this criterion and will qualify for the study.
   * Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Have previously received treatment with topoisomerase I inhibitors as a free form or as other formulations.
8. Have previously received treatment in advanced or metastatic setting with systemic therapy before or after the first line CDK4/6i combined with ET, including but not limited to:

   1. chemotherapy.
   2. endocrine monotherapy or combined with target therapy (PI3Ki, mTORi, AKTi, HDACi, etc.).
   3. PARPi.
   4. immune checkpoint inhibitors (PD-1, PD-L1, CTLA-4, etc.)
   5. antibody-drug conjugates.
9. Have an active second malignancy. Note: patients with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (e.g., nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
10. Met any of the following criteria for cardiac disease:

    1. Myocardial infarction or unstable angina pectoris within 6 months of enrollment.
    2. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
    3. New York Heart Association (NYHA) class III or greater congestive heart failure or left ventricular ejection fraction of < 40%.
11. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
12. Have active serious infection requiring antibiotics.
13. Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody, if done at screening) with detectable viral load OR taking medications that may interfere with SN-38 metabolism.
14. Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.

    * Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
    * Patients who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require an HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
    * Patients who test positive for HIV antibody.
15. Patients with a history of or current central nervous system (CNS) metastases. A scan to confirm the absence of brain metastases was not required. Patients with unknown CNS metastatic status and any clinical signs indicative of CNS metastases were eligible if CNS metastases were excluded using CT and/or MRI scans.
16. Patients with Gilberts disease.
17. Known history of clinically significant active chronic obstructive pulmonary disease, or other moderate-to-severe chronic respiratory illness present within 6 months of the first dose.
18. High-dose systemic corticosteroids within 2 weeks prior to the first dose (however, low-dose corticosteroids 10 mg prednisone or equivalent daily were permitted if provided the dose was stable for 4 weeks).
19. Scheduled surgery during the study, other than minor surgery which would not delay study treatment.
20. Patients who had received a live vaccine within 30 days of the first dose.
21. Rapid deterioration during Screening prior to the first dose, e.g., significant change in PS, unstable pain symptoms requiring modifications in analgesic management.
22. Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
23. Any medical condition that, in the investigators or sponsor's opinion, poses an undue risk to the patient's participation in the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year
  assessed by the incidence, nature, and severity of adverse events (AEs; NCI CTCAE v5.0)

SECONDARY OUTCOMES:
ORR | up to 16 weeks
  Objective Response Rate: Proportion of patients with a predefined tumor size reduction (Complete Response + Partial Response
DoR | From date of treatment initiation until the date of first documented progression, assessed up to 24 months
  Duration of Response: Time from first response (CR/PR) to disease progression or death
DCR | up to 24 weeks
  Disease Control Rate: Proportion of patients achieving CR, PR, or Stable Disease (SD)
PFS | From date of treatment initiation until the date of first documented progression or death from any cause, assessed up to 24 months
  Progression-Free Survival: Time from treatment initiation to disease progression or death
OS | From date of treatment initiation until the date of death from any cause, assessed up to 60 months
  Overall Survival: Time from treatment initiation to death from any cause
PROs | through study completion, an average of 1 year
  according to nine items subset derived from PRO-CTCAE® Item Library Version 1.0: decreased appetite, nausea, vomiting, constipation, diarrhea, pain in the abdomen, shortness of breath, hair loss, and fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China